CLINICAL TRIAL: NCT06558097
Title: A First-in-human, Randomized, Sponsor Open-label, Participant and Investigator Blinded, Placebo-controlled, Single Ascending Dose Study to Explore the Safety, Tolerability and Pharmacokinetics of XXB750 in Healthy Participants
Brief Title: Safety, Tolerability, and Pharmacokinetics of XXB750 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CXXB750A02101
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: XXB750 in Healthy Participants
Keywords: XXB750; healthy participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- XXB750 s.c 1 mg (Experimental): Single SC dose of XXB750 1 mg
  Interventions: Drug: XXB750
- XXB750 s.c 3 mg (Experimental): Single SC dose of XXB750 3 mg
  Interventions: Drug: XXB750
- XXB750 s.c 10 mg (Experimental): Single SC dose of XXB750 10 mg
  Interventions: Drug: XXB750
- XXB750 s.c 30 mg (Experimental): Single SC dose of XXB750 30 mg
  Interventions: Drug: XXB750
- XXB750 s.c 60 mg (Experimental): Single SC dose of XXB750 60 mg
  Interventions: Drug: XXB750
- XXB750 s.c 120 mg (Experimental): Single SC dose of XXB750 120 mg
  Interventions: Drug: XXB750
- XXB750 s.c 240 mg (Experimental): Single SC dose of XXB750 240 mg
  Interventions: Drug: XXB750
- Placebo (Placebo Comparator): Placebo to XXB750
  Interventions: Other: Placebo
- XXB750 s.c 240 mg Japanese cohort (Experimental): Single SC dose of XXB750 240 mg in the Japanese cohort
  Interventions: Drug: XXB750
- Placebo for Japanese cohort (Placebo Comparator): Placebo to XXB750 in the Japanese cohort
  Interventions: Other: Placebo
- XXB750 s.c 450 mg (HBP) (Experimental): Single SC dose of XXB750 450 mg (High Blood Pressure Cohort)
  Interventions: Drug: XXB750
- XXB750 s.c 600 mg (HBP) (Experimental): Single SC dose of XXB750 600 mg (High Blood Pressure Cohort)
  Interventions: Drug: XXB750
- Placebo to High Blood Pressure cohort (Placebo Comparator): Placebo to XXB750 in High Blood Pressure cohorts
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: XXB750 — Single SC dose of XXB750 (administered by single or multiple injections)
  Arms: XXB750 s.c 1 mg; XXB750 s.c 10 mg; XXB750 s.c 120 mg; XXB750 s.c 240 mg; XXB750 s.c 240 mg Japanese cohort; XXB750 s.c 3 mg; XXB750 s.c 30 mg; XXB750 s.c 450 mg (HBP); XXB750 s.c 60 mg; XXB750 s.c 600 mg (HBP)
Other: Placebo — Single SC dose of matching placebo (administered by single or multiple injections)
  Arms: Placebo; Placebo for Japanese cohort; Placebo to High Blood Pressure cohort

SUMMARY:
This study was a randomized, participant and investigator-blinded, placebo-controlled, single-ascending dose study, consisting of 9 sequential dose cohorts (1 mg, 3 mg, 10 mg, 30 mg, 60 mg, 120 mg, 240 mg, 450 mg and 600 mg) and a Japanese ethnic sensitivity cohort (240 mg dose)

DETAILED DESCRIPTION:
Eligible healthy participants with normal blood pressure (SBP: 110-139 mmHg; DBP: 70-89 mmHg) were randomized into dose cohorts 1 - 240 mg. Eligible healthy participants with elevated blood pressure (SBP: 139 - 159 mmHg; DBP: 75 - 95 mmHg) were randomized into dose cohorts 450 and 600 mg. Each participant received a subcutaneous single dose of either XXB750 or placebo. In total, the duration of the study was 151 days, including the full Screening period of up to 28 days, safety, pharmacokinetics and pharmacodynamics assessments over a period of 91 days, and a 30-day safety follow up call after the end of study visit.

Sentinel dosing will be applied in this FIH study at each new dose level to ensure participant's safety and minimize the number of participants that may experience symptomatic hypotension, especially for sustained periods of time attributing to the long acting nature of XXB750 and the sustained pharmacological effects on BP at higher doses. The 10-day safety monitoring for the sentinel cohort is considered sufficient based on the predicted mean Tmax (4.5 days) in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants age 18 to 50 years of age included, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Participants must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 32 kg/m2. BMI = Body weight (kg) / [Height (m)]2
* For ethnic Japanese cohort: participants must be defined as being of first, second or third generation ethnic origin, with each set of parents qualifying as Japanese under the prior generation.

Exclusion Criteria:

* Any surgical or medical condition which significantly altered the distribution, metabolism, or excretion of drugs, or which jeopardized the participant's participation in the study.
* Known history or current clinically significant arrhythmias.
* Women of child-bearing potential were excluded from this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | Up to 121 days
  To evaluate the safety and tolerability of single ascending SC doses of XXB750 in healthy participants.
  Adverse events may include abnormal vital signs, safety laboratory tests, physical exam tests and ECG parameters that include clinical signs or symptoms, are considered clinically significant or require therapy.

SECONDARY OUTCOMES:
Pharmacokinetics parameters: Tmax | Up to 91 days
  To evaluate the pharmacokinetics: Time to maximum concentation (Tmax) of XXB750 in healthy participants following a single SC dose of XXB750.
Pharmacokinetics parameters: Cmax | Up to 91 days
  To evaluate the pharmacokinetics: Peak plasma concentration (Cmax) of XXB750 in healthy participants following a single SC dose of XXB750.
Pharmacokinetics parameters: AUClast | Up to 91 days
  To evaluate the pharmacokinetics: Area under the plasma concentration curve (AUClast) of XXB750 in healthy participants following a single SC dose of XXB750.
Pharmacokinetics parameters: AUCinf | Up to 91 days
  To evaluate the pharmacokinetics: Area under the curve (AUCinf) of XXB750 in healthy participants following a single SC dose of XXB750.
Pharmacokinetics parameters: T1/2 | Up to 91 days
  To evaluate the pharmacokinetics: Half-life (T1/2) of XXB750 in healthy participants following a single SC dose of XXB750.
Pharmacokinetics parameters: Vz/F | Up to 91 days
  To evaluate the pharmacokinetics: Vd/F of XXB750 in healthy participants following a single SC dose of XXB750.
Pharmacokinetics parameters: CL/F | Up to 91 days
  To evaluate the pharmacokinetics: Apparent clearance (CL/F) of XXB750 in healthy participants following a single SC dose of XXB750.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No